CLINICAL TRIAL: NCT07340840
Title: THE RHYTHM OF CALM: EFFECTS OF RECREATIONAL YOGA ON EMOTIONAL AND AUTONOMIC HEALTH AMONG NURSING HOME RESIDENTS
Brief Title: Recreational Yoga and Emotional-Autonomic Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hüseyin Gümüş, Profesör, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU Ethics Committee 2023/020
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Depression in Older Adults; Heart Rate Variability (HRV)
Keywords: Yoga; Depression; Leisure; Heart rate variability; Nursing home
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recreational Yoga Intervention Group (Experimental): Participants in this group take part in a recreational therapy-based yoga program conducted twice weekly for 10 weeks. Each session lasts approximately 40-60 minutes and includes gentle yoga postures, breathing exercises, relaxation techniques, and meditation. The yoga program is designed to be safe and appropriate for older adults living in a nursing home and is supervised throughout the intervention period.
  Interventions: Behavioral: Recreational Therapy-Based Yoga
- Control Group (No Intervention): Participants in the control group do not receive any structured exercise or recreational intervention during the study period and continue their usual daily activities within the nursing home.

INTERVENTIONS:
Behavioral: Recreational Therapy-Based Yoga — The yoga intervention consists of supervised group sessions including relaxation exercises, basic and progressive yoga postures (asanas), breathing exercises, and meditation. Sessions are held twice per week for 10 weeks. Supportive equipment such as chairs, cushions, blocks, and towels is used to ensure participant comfort and minimize injury risk.
  Arms: Recreational Yoga Intervention Group

SUMMARY:
Older adults living in nursing homes often experience depression, reduced satisfaction with daily activities, and changes in heart rhythm related to the autonomic nervous system. Non-drug approaches that are safe and easy to apply may help improve both emotional well-being and physical health in this population.

This randomized controlled study investigates the effects of a recreational therapy-based yoga program on emotional health and autonomic nervous system function in nursing home residents aged 65 years and older. Participants are randomly assigned to either a yoga intervention group or a control group. The yoga group participates in supervised yoga sessions twice a week for 10 weeks, including gentle yoga postures, breathing exercises, relaxation, and meditation. The control group does not receive any structured intervention during the study period.

Depression levels, leisure time satisfaction, and heart rate variability are measured before and after the intervention. Heart rate variability is used as an indicator of autonomic nervous system regulation. The study aims to determine whether recreational yoga can be a safe, low-cost, and effective non-pharmacological approach to improve emotional well-being and autonomic health among older adults living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older.
* Living in a nursing home.
* Able to communicate and follow instructions.
* Voluntary participation with signed informed consent.
* Available to participate in the 10-week study protocol

Exclusion Criteria:

* Participation in therapy-based practices (e.g., yoga, reiki, massage) within the last month.
* Being bedridden.
* Use of psychiatric medications.
* Irregular participation in the 10-week yoga program.
* Failure to complete pre-test or post-test assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Depression Level | Baseline (pre-intervention) and immediately after the 10-week intervention period
  Depression levels are assessed using the Geriatric Depression Scale-15 (GDS-15), a validated self-report questionnaire for older adults. Higher scores indicate greater depressive symptoms.
Heart Rate Variability (HRV) | Baseline (pre-intervention) and immediately after the 10-week intervention period
  Autonomic nervous system function is evaluated using heart rate variability parameters measured with a chest-worn heart rate monitor. Time-domain, frequency-domain, and non-linear HRV parameters are analyzed to assess sympathetic and parasympathetic activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No